CLINICAL TRIAL: NCT05280054
Title: An Open-label, Drug Interaction Study to Evaluate Safety, Pharmacokinetic, and Pharmacodynamic Effect of Oral Administration of AV-101 Alone and in Combination With Probenecid in Healthy Subjects
Brief Title: AV-101 Alone and in Combination With Probenecid in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: VistaGen Therapeutics, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AV-101 CL005
Record Dates: First submitted 2021-12-27; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-12

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — 4-chlorokynurenine; Probenecid

STUDY DESIGN:
Intervention Model Description: AV-101 alone followed by AV-101 + Probenecid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AV-101 (Experimental): AV-101 360 mg oral capsules single dose
  Interventions: Drug: AV-101
- AV-101 + Probenecid (Experimental): AV-101 360 mg oral capsules + 1000 mg Probenecid
  Interventions: Drug: AV-101; Drug: Probenecid

INTERVENTIONS:
Drug: AV-101 — 360 mg capsules
  Other Names: 4-chloro-kynurenine
Drug: Probenecid — 1000 mg oral
  Arms: AV-101 + Probenecid

SUMMARY:
This is an open-label, two period, fixed-sequence, drug-drug interaction study to compare the PK and PD of orally administered AV-101 alone and in combination with probenecid in healthy subjects. In Treatment Period 1, subjects will receive AV-101 following an overnight fast of at least 8 hours. In Treatment Period 2, subjects will fast overnight for at least 8 hours, and then receive AV-101 2 hours after receiving 1,000 mg probenecid. Each Treatment Period will be separated by a washout period. The doses of AV-101 in Cohort 1 and a possible Cohort 2 will be 360 mg and 720 mg, respectively. Optional Cohorts 3 and 4 may be enrolled depending on results from Cohorts 1 and 2. CSF will be collected via indwelling catheter to determine the PK of AV-101 and its active metabolite 7-Cl-KYNA.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be a male or non-pregnant, non-breastfeeding female.
2. Subject must be between 18 and 55 years of age (inclusive) at the Screening Visit.
3. The subject has a body mass index (BMI) between 18.5 kg/m2 and 30 kg/m2 inclusive, with a minimal body weight of 60 kg.
4. Female subjects must agree to use double barrier contraception (condom for male partner) and the female using an acceptable form of birth control from screening until 14 days after completion of the study.
5. Subject is willing and able to remain in the clinic research unit for the entire duration of each confinement period.
6. Subject must be clinically healthy, as assessed by the Investigator, to participate in the study, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12-lead electrocardiogram (ECG), and vital sign measurements performed at the Screening Visit and Admission. Repeat assessment may be performed at the Screening Visit

Exclusion Criteria:

1. Subject on over-the-counter, herbal and prescription medications as well as investigational medicinal products (IMP)s and not completing 14 days or 5 half-lives whichever is longer at the time of screening should be excluded.
2. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
3. Has a clinically significant abnormal finding on the physical exam, medical history, ECG, or clinical laboratory results at screening that in the opinion of the Investigator would preclude the subject from safely participating in the trial.-
4. Is a female with a positive pregnancy test result.
5. Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, marijuana, methylenedioxymethamphetamine, oxycodone, phencyclidine, tricyclic antidepressants, propoxyphene, and opiates).
6. Has a positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or Human Immunodeficiency Virus (HIV) at screening or has been previously treated for Hepatitis B, Hepatitis C, or HIV infection.
7. Subject with a QT interval corrected for heart rate using Fridericia's correction (QTcF) greater than 450 ms (males) or greater than 470 ms (females), at screening obtained after at least 5 minutes rest in a supine position using the ECG machine algorithm.
8. Subject with a history of allergic reaction to probenecid.
9. History of suicide behavior and ideation. At screening, if the C-SSRS responses ("yes" answers to item 4 or 5) indicate that the subject may have experienced suicidal ideation associated with actual intent or plan within 12 months of screening, may have had a history of suicidal behavior within the past 10 years, or had any lifetime history of recurrent suicidal behavior, the subject will be excluded from participation in the study.
10. Subject who has a positive reverse transcription polymerase chain reaction (RT-PCR) test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2; coronavirus disease 2019 [COVID-19]) during the Screening or a positive Rapid Swab test for SARS-CoV-2 at Admission.
11. Subject who has clinical signs and symptoms consistent with SARS-CoV-2 infection, e.g., fever, dry cough, dyspnea, sore throat, fatigue, or positive SARS-CoV-2 test result within 14 days prior to the Screening Visit or at Admission.
12. Subject who had a severe course of SARS-CoV-2 (extracorporeal membrane oxygenation, mechanically ventilated).
13. Subject who has recent (within 14 days prior to the Screening Visit or between the Screening Visit and the Admission) exposure to someone who has SARS-CoV-2 symptoms or positive test result.
14. Hypersensitivity to anesthetic or derivatives used during CSF collection or any medication used to prepare the area of the lumbar puncture (LP).
15. Previous CSF collection within 30 days prior to admission (Day -1) to the clinic research unit.
16. History of vertebral deformities, major lumbar back surgery, clinically significant back pain, clinically significant abnormal X-ray, and/or injury, in the opinion of the Investigator that would preclude the subject participation or CSF collection during study not possible.
17. An ongoing skin infection at the LP site.
18. Clinically significant coagulation tests values outside the normal reference range (prothrombin time/international normalized ratio, partial thromboplastin time) at screening per Principal Investigator discretion.
19. Evidence of disease within 4 weeks before dosing related to chronic headache, migraines, joint pain or other disorders or disease resulting in chronic or intermittent pain.
20. Any personal or family history of seizure (including febrile seizures) or diagnosis of epilepsy or episode of unexplained loss of consciousness.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Plasma and CSF concentrations of 7-chloro-kynurenic acid (7-Cl-KYNA) in ng/ml | 24 hours
  Difference in 7-Cl-KYNA levels after AV-101 with and without probenecid
Plasma and CSF concentrations of 4-chloro-kynurenine (AV-101) in ng/ml | 24 hours
  Difference in 4-Cl-KYN levels after AV-101 with and without probenecid

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel Early Phase Clinical Unit, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No